CLINICAL TRIAL: NCT01882127
Title: Clinical Study on All-Trans Retinoic Acid (ATRA) Combining High-dose Dexamethasone Versus High-dose Dexamethasone Alone for Initial Treatment of Primary Immune Thrombocytopenia (ITP)
Brief Title: All-Trans Retinoic Acid (ATRA) Combining Dexamethasone Versus High-dose Dexamethasone for Initial Treatment of Primary Immune Thrombocytopenia (ITP)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No eligible patient was enrolled.
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITP-009
Record Dates: First submitted 2013-04-19; First posted 2013-06-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2013-06

CONDITIONS: Purpura; Idiopathic Thrombocytopenic Purpura
Keywords: Purpura; Idiopathic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura; Purpura, Thrombocytopenic, Idiopathic | interventions — Tretinoin; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose-DEX (Active Comparator): 40 patients are enrolled to take dexamethasone orally at a dose of 40 mg daily for 4 days
  Interventions: Drug: Dexamethasone
- ATRA & High dose-DEX (Experimental): 40 patients are enrolled to take Dexamethasone orally at 40mg a day for 4 days and all-trans retinoic acid at 10mg tablet every 8 hours a day for 12 consecutive weeks.
  Interventions: Drug: All-Trans Retinoid Acid(ATRA); Drug: Dexamethasone

INTERVENTIONS:
Drug: All-Trans Retinoid Acid(ATRA) — patients in ATRA&High dose-DEX group take All-Trans Retinoic Acid(orally,10mg every 8 hours a day for 12 consecutive weeks) in combination with dexamethasone(intravenously , 40mg/d for 4 consecutive days).
  Other Names: Acid, trans-Retinoic; trans Retinoic Acid; all-trans-Retinoic Acid; Acid, all-trans-Retinoic; all trans Retinoic Acid
  Arms: ATRA & High dose-DEX
Drug: Dexamethasone — Patients in High dose-DEX treatment group take dexamethasone( orally , 40mg daily for 4 days),patients in ATRA&High dose-DEX group take All-Trans Retinoic Acid(orally,10mg every 8 hours a day for 12 consecutive weeks) in combination with dexamethasone(intravenously , 40mg/d for 4 consecutive days).

SUMMARY:
The project was undertaking by Qilu Hospital of Shandong University in China. In order to report the efficacy and safety of All-Trans Retinoic Acid (ATRA) combining with High-dose Dexamethasone for the treatment of adults with primary immune thrombocytopenia (ITP), compared to conventional high-dose dexamethasone therapy.

DETAILED DESCRIPTION:
The investigators are undertaking a parallel group, randomised controlled trial of 80 primary ITP adult patients from Qilu Hospital of Shandong University in China. One part of the participants are randomly selected to receive All-Trans Retinoic Acid(10mg tablet by mouth every 8 hours a day for 12 consecutive weeks, combining with dexamethasone (given orally at a dose of 40 mg per day for 4 days, the others are selected to receive high-dose of dexamethasone treatment (given orally at a dose of 40 mg daily for 4 days). Patients were monitored every 1 to 3 days at the first two weeks and every 1 to 4 weeks afterwards for platelet counts, and were monitored every 1 month for transaminitis and other side effects

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for immune thrombocytopenia.
2. Untreated hospitalized patients, may be male or female, between the ages of 18 ~ 80 years.
3. To show a platelet count < 30×10^9/L, and with bleeding manifestations.
4. Eastern Cooperative Oncology Group（ECOG）performance status ≤ 2.
5. Willing and able to sign written informed consent

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit.
2. Received high-dose steroids or [2] intravenous immunoglobulin transfusion(IVIG)in the 3 weeks prior to the start of the study.
3. Current HIV infection or hepatitis B virus or hepatitis C virus infections. Severe medical condition (lung, hepatic or renal disorder) other than ITP. 4.Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)

5.Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period.

6.Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.

7.Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Platelet count | up to six months per subject
  The outcome should be classified into one of the following descriptions accordingly :
  1. CR. A complete response (CR) was defined as a sustained (≥ 3 months) platelet count ≥ 100×10^9/L.
  2. R. A response (R) was defined as a sustained (≥ 3 months) platelet count ≥ 30×10^9/L without recurrence of thrombocytopenia.
  3. NR.No response (NR) was defined as platelet count < 30 × 10^9/L or a less than two fold increase in platelet count from baseline or the presence of bleeding. Platelet count must be measured on two occasions more than a day apart.
  4. Relapse.A relapse was defined as platelet count falls below 30×10^9/L or bleeding accrues after achieving R or CR.

OTHER OUTCOMES:
Bleeding episodes | up to six months per subject

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, Dr, Principal Investigator — Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Background] Toth K, Sarang Z, Scholtz B, Brazda P, Ghyselinck N, Chambon P, Fesus L, Szondy Z. Retinoids enhance glucocorticoid-induced apoptosis of T cells by facilitating glucocorticoid receptor-mediated transcription. Cell Death Differ. 2011 May;18(5):783-92. doi: 10.1038/cdd.2010.136. Epub 2010 Nov 12. PMID 21072052
- [Background] Tancini G, Marchini S. Adriamycin plus cyclophosphamide in advanced bronchial carcinoma. Tumori. 1976 Jul-Aug;62(4):373-5. doi: 10.1177/030089167606200403. PMID 1020044
- [Background] Tosi P, Pellacani A, Visani G, Ottaviani E, Ronconi S, Zamagni E, Benni M, Cavo M, Tura S. In vitro treatment with retinoids decreases bcl-2 protein expression and enhances dexamethasone-induced cytotoxicity and apoptosis in multiple myeloma cells. Eur J Haematol. 1999 Mar;62(3):143-8. doi: 10.1111/j.1600-0609.1999.tb01736.x. PMID 10089890
- [Background] Chen YH, Desai P, Shiao RT, Lavelle D, Haleem A, Chen J. Inhibition of myeloma cell growth by dexamethasone and all-trans retinoic acid: synergy through modulation of interleukin-6 autocrine loop at multiple sites. Blood. 1996 Jan 1;87(1):314-23. PMID 8547658